CLINICAL TRIAL: NCT04099056
Title: Brain Stimulation Studies of Decision-making Using Repetitive Transcranial Magnetic Stimulation (rTMS) and Temporal Interference (TI)
Brief Title: Brain Stimulation and Decision-making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Treadway, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00110965; F31MH127911 (NIH); 2025P011706 (Other: Emory IRB)
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: Transcranial magnetic stimulation (TMS); Temporal Interference (TI)
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Participants with Major Depressive Disorder (MDD) (Active Comparator): Participants with MDD will complete computer tasks while receiving TMS/ TI
  Interventions: Device: Neurostimulation
- Healthy Control (Active Comparator): Participants without MDD will complete computer tasks while receiving TMS/TI
  Interventions: Device: Neurostimulation

INTERVENTIONS:
Device: Neurostimulation — Participants will be seated comfortably in a chair and asked to complete simple computer tasks. Participants will receive neurostimulation in the form of Transcranial Magnetic Stimulation (TMS) or Temporal Interference (TI).
  TMS: Either during, or just before any of the tasks, participants will receive either repetitive transcranial magnetic stimulation (rTMS) or single pulse TMS. During this, the researchers place a small plastic coil next to the participant's head. The coil will then generate a magnetic pulse, and stimulation will occur during presentation of the visual stimuli on which subjects will conduct behavioral or cognitive tasks.
  TI: Either during, or just before, any of the above tasks, participants will receive stimulation with TI. To do so, commercially available gel-based electrodes will be placed on the scalp to target the relevant brain region. The position targeted by the electrodes will be guided by previously defined coordinates.

SUMMARY:
Decision-making is an important process that is frequently shown to be impaired in patients with depression. While a number of preclinical and clinical studies have identified key regions involved in this process, it remains unclear exactly how these regions are influencing choice behavior especially when choices become more challenging. The goal of this project is to understand how these regions, such as the cingulate cortex, impact difficult choice behavior. Specifically, the researchers are interested in learning how disruptions in cognitive control might impact choice preferences during difficult decisions in depressed patients. To do this, this study will recruit participants with depression (as well as healthy controls) to perform game-like tasks in the laboratory while undergoing TMS or TI.

DETAILED DESCRIPTION:
In recent years, countless studies have employed functional magnetic resonance imaging (fMRI) and other imaging modalities to both discover and track activity in brain regions involved in performance or behavior in a wide range of tasks. Running in parallel, research involving neuromodulation has afforded researchers the opportunity to test the impact of direct stimulation on areas hypothesized to be involved in certain processes or behaviors. Among such technologies are transcranial magnetic stimulation (TMS) and temporal interference (TI).

TMS and TI can be performed during any sort of cognitive or behavioral task to estimate the effect of the stimulated brain area; as such, TMS and TI have an exciting array of potential applications in research. One area, for example, is cost-benefit decision-making. Because of the potential biases associated with self-report measures-including simple recall errors, misinterpretations of the item, and social-conformity pressures-a number of psychological laboratories have advocated for the use of decision-making tasks as an alternative means of assessing motivation and reward-related symptoms. Such tasks ask individuals to choose how much they are willing to work, wait, or risk to win various rewards. These measures have been used in a variety of behavioral and neuroimaging studies and in different clinical populations.

This study will use TMS or TI in combination with a series of behavioral tasks to probe the relationship between areas known or hypothesized to be involved in cognition and/or cost-benefit decision-making, and performance on these tasks. This study aims to understand the effect of TMS or TI stimulation of certain brain areas on performance in a series of cognition- and decision-based behavioral tasks. To do so, the researchers will stimulate areas of the cortex hypothesized to be selectively engaged with cognition of a given category, or cost-benefit decision-making (depending on the behavioral tasks used). This study will examine healthy controls and depressed patients to investigate these effects. Such an aim will not only provide a deeper understanding of decision-making for basic research but will also hopefully inform understanding when decision-making is altered, as in psychiatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* Fluent English speaker
* Absence of current drug use as assessed by subject history and/or urine drug screen

Exclusion Criteria:

* Pregnant or currently breastfeeding women or any woman of childbearing potential who is seeking to become pregnant or suspects that she may be pregnant, as assessed by subject report and/or urine pregnancy screen
* Contraindications to fMRI scanning (including presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia) as assessed with the standard MRI screening form from the Facility for Research and Education in Neuroscience (FERN)
* Unable to fit comfortably in the scanner
* Contraindication to TMS, including history or family history of epilepsy, metallic implants in the head and/or neck, brain stimulators, vagus nerve stimulators, ventriculoperitoneal (VP) shunt, pacemakers
* Current use of medications that may increase the risk of seizures (e.g., bupropion, varenicline, chlorpromazine, theophylline) or reduce the effects of rTMS, such as benzodiazepines
* History or current serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic disease, as assessed by subject history
* Not right-handed as assessed by the Chapman handedness inventory or self-report
* History of head injury resulting in more than a brief loss of consciousness, as assessed by subject history
* History of cocaine or stimulant use (e.g., amphetamine, cocaine, methamphetamine), as assessed by subject history
* History of use of dopaminergic drugs (including methylphenidate or other stimulant medication), as assessed by subject history
* Current use or more than occasional use in the past year of tobacco products, including cigarettes, e-cigarettes, cigars, snuff, and chewing tobacco, or nicotine replacement products such as gum or patches, as assessed by subject history
* Evidence of significant inconsistencies in self-report measures

Additional Exclusion Criteria for Optional Ecological Momentary Assessment (EMA)Component for Subject Safety

* Anything above minimal risk for suicide, as assessed during the clinical interview (SCID) at screening and the Columbia Suicide Severity Rating Scale (C-SSR). C-SSRS risk will be assessed as any score > 3.
* Any physical or neuropsychiatric conditions that may worsen/or prevent walking or running.

Additional Exclusion Criteria for Optional Ecological Momentary Assessment (EMA)Component for Data Quality

* Meet criteria for current psychotic disorders, bipolar disorders, or severe substance use disorders as assessed by the Mini International Neuropsychiatric Interview.
* Used psychotropic medications within the last six weeks as assessed by subject history.

Additional Exclusion Criteria for Participants with Major Depressive Disorder:

* Anything above minimal risk for suicide, as assessed during the clinical interview (SCID) at screening and the Columbia Suicide Severity Rating Scale (C-SSRS)
* A symptom severity score of at least 11, as assessed by the Beck Depression Inventory (BDI)-II
* History or current diagnosis of any of the following Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV psychiatric illnesses:

  * Organic mental disorder
  * Schizophrenia spectrum disorders
  * Delusional disorder
  * Psychotic disorders not otherwise specified
  * Patients with mood-congruent or mood-incongruent psychotic features
  * Patients with bipolar mood disorders
  * Substance dependence
  * Substance abuse within the last 12 months (except cocaine or stimulant abuse), which will lead to exclusion
* Absence of any psychotropic medications for at least 2 weeks. No patient will be asked to discontinue or otherwise interrupt any psychotropic medications to participate in this study. The listed "washout" periods are only applicable for patients who previously used psychotropic medications, but recently decided to discontinue their use for some other reason.

  * 6 weeks for fluoxetine
  * 6 months for neuroleptics
  * 2 weeks for benzodiazepines
  * 2 weeks for any other antidepressants

Additional Exclusion Criteria for Healthy Controls:

* Any current or past history of any DSM-IV psychiatric illnesses, presence of a DSM-IV psychiatric disorder within a first-degree relative, or current or past use of psychotropic medications
* Score no greater than 10 on the BDI-II
* Score > 1 on the SHAPS

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Staggered Effort-Based Decision-Making Task | Day 1, during TMS/ TI stimulation
  Assessment of reward motivation will be accomplished using an effort-based decision-making task modified for fMRI use. During each trial, subjects are presented with a choice between two levels of task difficulty, a High Effort option and a Low Effort option, which require different amounts of speeded manual button pressing for differing levels of monetary reward. The reward magnitude for a No Effort option remains constant ($1.00), while the reward magnitude for the High Effort option varies from $1.00 to $11.00. Additionally, the amount of effort required for the High Effort option will vary between 20%, 50%, 80% and 100% of the subject's max effort (set for each individual prior to scan). Multiple metrics of task performance will be compared between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Treadway, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No